CLINICAL TRIAL: NCT02045758
Title: A Study to Compare Analyte Levels in Blood Samples Collected Using the TAP20-C Device With Results Obtained by Fingerstick
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seventh Sense Biosystems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-P002
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP20-C (Experimental): TAP20-C
  Interventions: Device: TAP20-C
- Fingerstick (Active Comparator): Fingerstick
  Interventions: Device: Fingerstick

INTERVENTIONS:
Device: Fingerstick
  Arms: Fingerstick
Device: TAP20-C
  Arms: TAP20-C

SUMMARY:
This study will compare blood collection from the forearm using an investigational device TAP20-C to blood collection from the fingertip.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subject Group

  1. Male and female volunteers 18 years of age or older.
  2. Voluntary written consent to participate in this study. Diabetic Subject Group

  <!-- -->

  1. Male and female volunteers 18 years of age or older.
  2. Have been diagnosed with Type 1 or Type 2 diabetes mellitus by self-report.
  3. Voluntary written consent to participate in this study.

Exclusion Criteria:

1. Subjects who are pregnant or nursing mothers by self-report.
2. Subjects with a history of skin disorders or who present with abnormal skin integrity or atypical skin health within the areas to be tested.
3. Subjects with a missing index or middle finger on either hand or a missing forearm
4. Subjects who have known allergies to titanium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Non-Inferiority of Analyte Levels | Day 1
  The study will compare the concentrations of various analytes in blood samples collected by both collection methods in a single 2 hour session.

CONTACTS AND LOCATIONS:
Locations (1):
- Seventh Sense Biosystems, Cambridge, Massachusetts, United States